CLINICAL TRIAL: NCT05191446
Title: Impact of the Coronavirus 2019 (COVID-19) Pandemic on Patient Outcomes, Telehealth Care Delivery, and Treatment for Unhealthy Alcohol Use in Vulnerable Patients With Advanced Liver Disease Across Two Healthcare Systems
Brief Title: Coronavirus Disease 2019 (Covid-19) Impact on Alcohol-related Liver Disease Patient Outcomes, Care and Alcohol Use
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-33076; R01AA029312 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-01-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Liver Diseases; Alcohol Use Disorder
MeSH Terms: conditions — Liver Diseases; Alcoholism | interventions — Ethanol; Methods; diamine N-acetyltransferase

STUDY DESIGN:
Intervention Model Description: Randomized trial with patients assigned to an experimental condition or to usual care.
Who Masked: Outcomes Assessor
Masking Description: Research assistants completing follow up interviews with participants will be blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped alcohol intervention (SAT) to reduce unhealthy alcohol use (Experimental): For participants randomized to SAT, consistent with stepped care, treatment will begin with lower intensity services that are stepped up, if necessary, at a predefined time point. Step 1 consists of three motivational interviewing (MI)sessions delivered every 2 weeks. At the 3-month assessment, those with non-response to MI, defined as continued unhealthy alcohol use in the prior 14 days, will be referred to on site physician managed addiction specialty services (Step 2) for higher intensity services.
  Interventions: Behavioral: Stepped alcohol intervention (SAT) to reduce unhealthy alcohol use
- Usual Care (UC) (Active Comparator): UC participants will receive their usual services in hepatology. They will also be given publicly available patient education materials regarding risk associated with unhealthy drinking (mail/email or in-person if desired) and will be asked to follow up with their physician should they have questions about information provided in the handouts. UC participants' hepatology provider will be notified if AUDIT-C scores are greater than 3 at baseline. All UC participants will have access to alcohol and other substance use treatment available to patients at their respective sites.
  Interventions: Other: Usual Care (UC)

INTERVENTIONS:
Behavioral: Stepped alcohol intervention (SAT) to reduce unhealthy alcohol use — Step 1 includes three sessions of motivational interviewing (MI). MI will consist of three video (Zoom) or telephone sessions: an initial 45-minute session, followed by two 20-minute sessions. Treatment is based on "Motivational Interviewing" by Miller and Rollnick, and includes exploring ambivalence about change, reflective listening, expressing empathy, and discussion about change. To support increased motivation to reduce drinking, discussion will center on effects of hazardous drinking on liver disease.
  Step 2 includes referral to addiction medicine for participants who do not reduce unhealthy alcohol use or requested by patient. Specialty addiction services include both direct treatment and coordination of addiction care. After an evaluation, the addiction medicine physician may recommend pharmacotherapy (in consultation with hepatology provider if indicated), and/or referral to intensive outpatient, or residential level of care depending on clinical judgement.
  Arms: Stepped alcohol intervention (SAT) to reduce unhealthy alcohol use
Other: Usual Care (UC) — UC participants will receive their usual services in hepatology. They will also be given publicly available patient education materials regarding risk associated with unhealthy drinking (mail/email or in-person if desired) and will be asked to follow up with their physician should they have questions about information provided in the handouts. UC participants' hepatology provider will be notified if AUDIT-C scores are greater than 3 at baseline. All UC participants will have access to alcohol and other substance use treatment available to patients at their respective sites.
  Arms: Usual Care (UC)

SUMMARY:
The study consists of a randomized controlled trial evaluating the efficacy and feasibility of a stepped alcohol treatment using telemedicine on unhealthy alcohol use in patients with chronic liver disease receiving care in hepatology practices at three sites. Patients who meet eligibility criteria will be randomized to one of two study arms: 1) Stepped Alcohol Treatment (SAT) or, 2) Usual Care (UC). Participants will be randomized separately by site. SAT includes 3 sessions of motivational interviewing followed by referral to addiction medicine for patients who do not reduce unhealthy drinking. Trial outcome measures will be complete at 6 and 12 months following baseline enrollment.

DETAILED DESCRIPTION:
Background/Rationale: Unhealthy alcohol use is consumption of alcohol at more than the "moderate" levels of up to 1 drink per day (7/week) for women and up to 2 drinks per day (14/week) for men, as defined by NIAAA. Unhealthy alcohol use is prevalent in chronic liver disease (CLD), and for many patients no level of alcohol could be considered safe. Guidelines recommend integrated multidisciplinary care, but evidence-based strategies to address alcohol use beyond brief counseling are rarely provided in hepatology practices. A recent study showed that most veterans with cirrhosis and coexisting AUD do not receive behavioral treatment or pharmacotherapy for AUD. Similarly, in a study of cirrhosis patients [~70% alcohol-associated liver disease (ALD)] hospitalized at 4 safety net hospitals, less than half reported abstinence from alcohol, while 39% reported daily alcohol use, and alcoholic hepatitis accounted for the highest in-hospital mortality compared to other comorbidities. The investigators are focusing on these important outcomes in this study. Current guidelines recommend that brief intervention, pharmacotherapy, and referral to treatment should be offered to patients with ALD including those with alcohol use disorder (AUD) or advanced CLD of any etiology who drink alcohol at more than moderate amounts. Our approach follows these guidelines.

Overall approach: The investigators will enroll a total of 180 patients (90 assigned to stepped care, 90 to usual care) with liver disease and alcohol use; 60 patients will be recruited from each of the three study sites (two Veterans Administrations Healthcare System sites in Palo Alto and San Francisco as well as a safety net public clinic in San Francisco, CA). This intent-to-treat outcome study will include all patients recruited, whether or not they complete the interventions.

Recruitment: Hepatology practices at all three sites routinely screen patients for alcohol use. Eligible patients will be identified using the electronic medical record and, following permission from their provider, patients will be contacted about the study. Patients may also be referred directly by their hepatology providers. Interested patients who meet all eligibility criteria will be consented to participate in the study. The investigators will include English and Spanish speakers using bicultural and bilingual clinical research coordinators. Following enrollment, participants will have baseline, 3-, 6-, and 12-month assessments. Participants will be offered $50 for completing the baseline, 3-, and 6-month, and $100 for 12-month assessments.

Baseline assessment: At baseline, patient demographics (age, sex, race/ethnicity, income, education, insurance), medical history, medications, etiology of CLD, presence of cirrhosis or hepatic decompensation, history of illicit drugs, laboratory tests of liver function and COVID-19 will be captured using the electronic medical record. Measures of alcohol use will be performed using validated measures. Patients will then undergo randomization.

Randomization to study arms: Patients who meet study criteria will be randomized to one of two study arms: 1) Stepped Alcohol Treatment (SAT) or, 2) Usual Care (UC). See "Arms and Interventions" section for details.

Follow-up Assessments: A research staff member not participating in patient care will conduct follow-up interviews. He/she will be blinded to participants' treatment condition. Participants will be contacted by telephone at 3, 6 and 12 months to complete the measures. Patient reporting via telephone follow-up has been reliable in prior studies but a biomarker of alcohol use will also be performed to validate reports of alcohol abstinence

Statistical analysis: Repeated measures analyses will be conducted within a generalized linear mixed model (GLMM) framework. These models accommodate the range of continuous, count, and discrete outcomes that will be measured. Analyses will include treatment condition (SAT vs UC) as a between-subjects effect. Time (baseline, 3-month, 6-month, and 12-months) will be a repeated effect and the treatment x time interaction will be examined. Analyses will account for clustering of patients within study site.

Sample size: Sample size was determined using data from prior studies of MI and stepped care interventions for unhealthy alcohol use in individuals with liver disease and other populations, for the primary outcome (less than moderate alcohol use) and the secondary outcome of drinks per week.

Anticipated results: The investigators anticipate that SAT participants will be more likely than UC to reduce or be abstinent from alcohol use at the 3-, 6- and 12-month follow-up. The investigators also anticipate that SAT participants will have better clinical outcomes (less new or worsening clinical decompensation or hospitalizations) than controls at follow-up. The investigators will also explore COVID-19 related outcomes in both arms, e.g., infection rates, hospitalization and clinical outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Men and women age ≥ 18 years.
2. Diagnosis of chronic liver disease (CLD).
3. Unhealthy alcohol use, defined as more than moderate amount of alcohol use within the prior 30 days by National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria defined as on average more than 1 drink/day (7 drinks per week) for women and more than 2 drinks per day (14 drinks per week) for men, or on average at least one heavy drinking day (4+ drinks in a day for women and 5+ for men) per week in the prior 30 days. A standard drink is ~14 g of alcohol.
4. Ability to access a telephone or a digital device (i.e., computer, tablet or smart phone).

Exclusion criteria:

1. Severe medical or psychiatric conditions or evidence of acute alcohol intoxication preventing participation in the study
2. Are currently enrolled in formal treatment for unhealthy alcohol use, excluding self or mutual-help groups (e.g., Alcoholics Anonymous).
3. Women who are pregnant or breastfeeding or unwilling to use birth control.
4. Language preference other than English, Spanish or Chinese.
5. Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol use | 6 months after enrollment
  Less than moderate alcohol use in the prior 30 days at month 6 follow-up. Alcohol use survey questions will assess usual drinking frequency (days per week) and typical number of standard drinks consumed, in order to compute average number of drinks per week; and number of days of hazardous drinking (5+ drinks for men and, and 4+ drinks per women) in the past 30 days, using the Timeline Followback Method.

SECONDARY OUTCOMES:
Alcohol use cessation | 6 and 12 months after enrollment
  Alcohol use will be assessed at 6 months and 12 months following enrollment, using the Timeline Followback Method.
Drinks per week | 6 and 12 months after enrollment
  Alcohol use will be assessed at 6 months and 12 months following enrollment, using the Timeline Followback Method.
Liver-related outcomes | 6 and 12 months after enrollment
  Worsening liver function tests, new or worsening hepatic decompensation or new diagnosis of cirrhosis in those without advanced CLD, number of hospitalizations, Child-Pugh (A, B, and C) and Model of End stage Liver Disease (MELD) labs will be captured using electronic medical record data.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Khalili, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of california San Francisco, San Francisco, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
The study will comply with NOT-AA-19-020, "Notice of NIAAA Data-Sharing Policy for Human Subjects Grants Research Funded by the National Institute on Alcohol Abuse and Alcoholism (NIAAA)." NIAAA requires studies that include human subjects to submit de-identified data into the NIAAA data repository (NIAAADA), a NIAAA data repository hosted and managed by the National Institute of Mental Health (NIMH) Data Archive (NDA), in order to enable widespread data sharing. Key measurement domains include quality of life, patient satisfaction with care, use of telemedicine, health literacy measures, alcohol use, anxiety, depression, and use of health services. The investigators will obtain Informed Consent that allows for broad sharing of the research subjects' de-identified data and will follow all other necessary procedures as described in our Data Sharing and Archiving Plan.
Supporting Information: Study Protocol
Time Frame: The study team will submit data on or before the NDA submission due dates (April 1 and October 1 each year) in accordance with the applicable Data Sharing Terms and Conditions of award. The team will perform quality assurance (QA)/quality control (QC) checks on data within 4 months after the submission due dates and address any issues identified by the NDA. The study team will run the required NIAAADA data validation tool at least one time per month once data collection begins. Duration of availability will follow NIAAADA criteria.
Access Criteria: Access criteria will follow NIAAADA guidelines. The study team will Share data in accordance with the default NIAAADA data sharing schedule in accordance with the applicable Data Sharing Terms and Conditions of award.

REFERENCES:
- [Result] Satre DD, Dasarathy D, Batki SL, Ostacher MJ, Snyder HR, Hua W, Parekh P, Shui AM, Cheung R, Monto A, Wong RJ, Chen JY, Liao M, Tana M, Chen PH, Haight CG, Fakadej T, Khalili M. Factors Associated With Motivation to Reduce Alcohol Use Among Patients With Chronic Liver Disease. Aliment Pharmacol Ther. 2025 Feb;61(3):481-490. doi: 10.1111/apt.18387. Epub 2024 Nov 11. PMID 39523996
- [Result] Luk JW, Ha NB, Shui AM, Snyder HR, Batki SL, Ostacher MJ, Monto A, Wong RJ, Cheung R, Parekh P, Hua W, Tompkins DA, Fakadej T, Haight CG, Liao M, Khalili M, Satre DD. Demographic and clinical characteristics associated with utilization of alcohol use disorder treatment in a multicenter study of patients with alcohol-associated cirrhosis. Alcohol Clin Exp Res (Hoboken). 2025 Jan;49(1):244-255. doi: 10.1111/acer.15500. Epub 2024 Dec 4. PMID 39632077
- [Result] Wong RJ, Yang Z, Ostacher M, Zhang W, Satre D, Monto A, Khalili M, Singal AK, Cheung R. Alcohol Use Patterns During and After the COVID-19 Pandemic Among Veterans in the United States. Am J Med. 2024 Mar;137(3):236-239.e2. doi: 10.1016/j.amjmed.2023.11.013. Epub 2023 Dec 3. PMID 38052382
- [Result] Athavale P, Wong RJ, Satre DD, Monto A, Cheung R, Chen JY, Batki SL, Ostacher MJ, Snyder HR, Widiarto BD, Oh SY, Liao M, Viviani AML, Khalili M. Telehepatology Use and Satisfaction Among Vulnerable Cirrhosis Patients Across Three Healthcare Systems in the Coronavirus Disease Pandemic Era. Gastro Hep Adv. 2023 Nov 20;3(2):201-209. doi: 10.1016/j.gastha.2023.11.006. eCollection 2024. PMID 39129958
- [Result] Luk JW, Satre DD, Cheung R, Wong RJ, Monto A, Chen JY, Batki SL, Ostacher MJ, Snyder HR, Shui AM, Liao M, Haight CG, Khalili M. Problematic alcohol use and its impact on liver disease quality of life in a multicenter study of patients with cirrhosis. Hepatol Commun. 2024 Feb 3;8(2):e0379. doi: 10.1097/HC9.0000000000000379. eCollection 2024 Feb 1. PMID 38315141
- [Result] Kim RG, Patel S, Satre DD, Shumway M, Chen JY, Magee C, Wong RJ, Monto A, Cheung R, Khalili M. Telehepatology Satisfaction Is Associated with Ethnicity: The Real-World Experience of a Vulnerable Population with Fatty Liver Disease. Dig Dis Sci. 2024 Mar;69(3):732-742. doi: 10.1007/s10620-023-08222-7. Epub 2024 Jan 13. PMID 38217682